CLINICAL TRIAL: NCT06412614
Title: Phenotypic Evaluation of Patients With Systemic Sclerosis Without Specific or Associated Autoantibodies
Brief Title: Evaluation of Patients With Systemic Sclerosis Without Specific or Associated Autoantibodies
Acronym: SCLERONAB
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI015
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SSc patients without specific or associated autoantibodies ("seronegative" patients)
  Interventions: Other: disease phenotype
- SSc patients with specific or associated autoantibodies
  Interventions: Other: disease phenotype

INTERVENTIONS:
Other: disease phenotype — evaluation of SSc phenotypes

SUMMARY:
Systemic sclerosis (SSc) is a complex systemic autoimmune disease with variable phenotype and prognosis. Autoantibodies are important diagnostic biomarkers in SSc. More than 90% of patients with SSc had anti-nuclear antibodies. Autoantibodies specific to SSc (anti-topoisomerase I antibodies, anti-centromeres, anti-RNA polymerase III, anti-Th/To, anti-fibrillarin, anti-NOR90) or associated with overlap syndromes (anti-RNA polymerase III antibodies -PM/Scl, anti-KU, anti-U1RNP, anti-TRIM21) are detected in most patients. Excluding anti-TRIM21 antibodies, autoantibodies are usually mutually exclusive and are associated with distinct phenotypes.

Around 5 to 10% of patients with SSc have no autoantibodies detectable with routine biological tests. Recently, new autoantibody specificities have been described in SSc (anti-eIF2B, anti-RuvBL1/2, anti-BICD2, anti-U11/U12 RNP antibodies).

"Seronegative" patients could represent new specificities of autoantibodies (unknown or not currently routinely evaluated) associated with different phenotypes of the disease.

Primary objective is to compare the phenotype of patients with systemic sclerosis with or without detectable specific or associated autoantibodies.

Secondary objectives are:

* to determine homogeneous groups of patients with systemic sclerosis without detectable specific or associated autoantibodies
* to compare the phenotype of patients with systemic sclerosis without detectable specific or associated autoantibodies according to anti-nuclear antibodies status

ELIGIBILITY:
Inclusion Criteria:

* Patient with systemic sclerosis defined according to ACR/EULAR 2013 classification criteria
* Patient with a minimum follow-up of 3 years since the diagnosis of systemic sclerosis
* Patient evaluated for the following systemic sclerosis specific and/or associated autoantibodies: anti-topoisomerase I, anti-centromere, anti-RNA polymerase III (RP155 and RP11), anti-Th/To antibodies , anti-fibrillarin, anti-NOR90, anti-PM/Scl, anti-KU, anti-U1RNP and anti-SSA antibodies (independently of antinuclear antibodies status)

Exclusion Criteria:

* Patient with equivocal results for one or more systemic sclerosis specific and/or associated autoantibodies
* Patient initially negative but with a positive result for systemic sclerosis specific and/or associated autoantibodies during follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in internal medicine or rheumatology units until December 2021
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2025-06-29 (Estimated); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
diagnosis time | baseline (J0)
  duration between date of first symptom (excluding Raynaud's phenomenon) and SSc diagnosis

SECONDARY OUTCOMES:
number of patients with scleroderma | baseline (J0)
  sine scleroderma (no scleroderma), limited scleroderma or diffuse scleroderma
number of patients with raynaud's phenomenon | baseline (J0)
number of patients with digital ulcers | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with calcinosis | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with telangiectases | baseline (J0)
number of patients with articular involvement | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with muscular involvement | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with cardiac involvement | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with interstitial lung disease | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with pulmonary arterial hypertension | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with scleroderma renal crisis | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
number of patients with gastrointestinal involvement | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
modified Rodnan skin score | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
forced vital capacity (FVC) | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
  %predicted FVC values
diffusing capacity for carbon monoxide (DLCO) | baseline (J0), 3 years of follow-up and through study completion (an average of 5 years)
  %predicted DLCO values
rate of patients without death | 3 years and 5 years of follow-up

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CH Dunkerque, Dunkirk
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU Nice, Nice
  - APHP, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No